CLINICAL TRIAL: NCT01682694
Title: Glucosamine and Chondroitin Effects
Acronym: GLANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 7798
Record Dates: First submitted 2012-09-04; First posted 2012-09-11 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Glucosamine; Chondroitin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucosamine and Chondroitin (Experimental): Glucosamine and Chondroitin
  Interventions: Dietary Supplement: Glucosamine and Chondroitin
- Placebo (Placebo Comparator): Inactive ingredients
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Glucosamine and Chondroitin — Glucosamine (1500 mg) and Chondroitin (1200 mg)
  Other Names: Nutramax
  Arms: Glucosamine and Chondroitin
Dietary Supplement: placebo
  Arms: Placebo

SUMMARY:
A common starting dose of glucosamine and chondroitin will reduce inflammation as reflected by a reduction in serum C-reactive protein.

DETAILED DESCRIPTION:
Use of glucosamine and chondroitin have been associated with reduced cancer and overall mortality. The aim of this study is to determine whether a common starting dose of glucosamine and chondroitin (1500 mg/d + 1200 mg/d, respectively) reduces systemic inflammation as reflected by a reduction in high sensitivity C-reactive protein.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Overweight (body mass index kg/m2 (BMI) between 25 and 32.5)
* Non-smoking men and women
* Aged 20-55y

Exclusion Criteria:

* Chronic medical illness, history of gastrointestinal, hepatic, or renal disorders, or inflammatory conditions (including autoimmune and inflammatory diseases)
* Pregnancy or lactation
* Currently on a weight-loss diet
* BMI (body mass index) < 25 or > 30
* Alcohol intake of greater than 2 drinks/day
* Current use of prescription or over-the-counter medications, (Excluding oral contraceptives and hormone-secreting IUDs), including use of aspirin or NSAIDs more than 2 days per week
* Abnormal renal, liver or metabolic test
* Inability to swallow pills
* Known allergy to shellfish
* Not willing to take pills made from shellfish or animal sources
* Intention to relocate out of study area within next 4 months

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
hsCRP | 1 year
  hsCRP is a biomarker of systemic inflammation

SECONDARY OUTCOMES:
untargeted (exploratory) serum metabolomics (differences in small molecule abundance ratios) | 1 year
  The mechanisms of action of glucosamine and chondroitin are currently unknown. Untargeted metabolomic assays of serum will be undertaken for exploratory analyses of potential effects of glucosamine and chondroitin. Significant differences in abundance ratios of small molecules between the intervention and placebo will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Navarro SL, White E, Kantor ED, Zhang Y, Rho J, Song X, Milne GL, Lampe PD, Lampe JW. Randomized trial of glucosamine and chondroitin supplementation on inflammation and oxidative stress biomarkers and plasma proteomics profiles in healthy humans. PLoS One. 2015 Feb 26;10(2):e0117534. doi: 10.1371/journal.pone.0117534. eCollection 2015. PMID 25719429